CLINICAL TRIAL: NCT06872385
Title: Profile of Brazilian Climacteric Women: the Brazilian Menopause Study
Acronym: Brazmenos
Status: Completed | Type: Observational
Sponsor: Faculdade de Medicina do ABC (Other)
Responsible Party: Principal Investigator, Luciano de Melo Pompei', Auxiliary Professor at Gynecology Department, Faculdade de Medicina do ABC
Other Study IDs: 24440719.0.0000.0082
Record Dates: First submitted 2022-01-20; First posted 2025-03-12 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Menopause
Keywords: menopause; hormone replacement therapy; epidemiology; knowledge

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Subjects: Women who meet the inclusion criteria and answered the questionnaire
  Interventions: Other: Answering a questionnaire

INTERVENTIONS:
Other: Answering a questionnaire — The subject have to answer an online questionnaire about her perceptions on menopause and opinion on treatments for the condition

SUMMARY:
Cross-sectional study with 1,500 women between 45 and 65 years old. Women participate by answering questionnaires prepared to get information about their perceptions and knowledge about menopause, hormone therapy and other treatments for menopause.

DETAILED DESCRIPTION:
This is a cross-sectional study with 1,500 women between 45 and 65 years old. The subjects participate by answering online questionnaires prepared to get information about their perceptions and knowledge about menopause, hormone therapy and other treatments for menopause. The distribution of subjects respect the distribution of Brazilian population according to country regions and according to socioeconomic class, and taking into account the information of last official Brazilian demographic census.

ELIGIBILITY:
Inclusion Criteria:

* Women between 45 and 65 years of age
* Women able to participate in a questionnaire on a digital platform and who have a device allowing this access

Exclusion Criteria:

* Pregnant or lactating women

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women aged between 45 and 65 years who accept to answer an online questionnaire in order to known their opinions on menopause and treatments for menopause, specially hormone therapy
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Actual)
Dates: Start 2019-11-29 (Actual); Primary Completion 2020-02-11 (Actual); Study Completion 2020-02-11 (Actual)

PRIMARY OUTCOMES:
Answer to the questionnaire | Day 1
  Subject has to answer the questionnaire with several questions about her heath condition, age at menopause, treatments used for menopause

CONTACTS AND LOCATIONS:
Overall Officials: Luciano M Pompei, Principal Investigator — Faculdade de Medicina do ABC
Locations (1):
- Faculdade de Medicina do ABC, Santo André, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided